CLINICAL TRIAL: NCT07043270
Title: 24BRO681 : Neoadjuvant Therapy With Alternating Gemcitabine Plus Nab-Paclitaxel and mFOLFIRINOX for Borderline Resectable Pancreatic Adenocarcinoma: A Phase 2 Clinical Trial
Brief Title: 24BRO681 : Alternating Gnp and mFOLFIRINOX for BR-PDAC
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Gabriel A. Brooks, Principal Investigator, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02002681; 24BRO681 (Other: DHMC); NCI-2022-08163 (Other: National Cancer Institute)
Record Dates: First submitted 2025-06-12; First posted 2025-06-29 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-05

CONDITIONS: Pancreas Adenocarcinoma
Keywords: mFOLFIRINOX; Gemcitabine; Nab-Paclitaxel; Neoadjuvant alternating chemotherapy; Resectable Pancreatic cancer; BR-PDAC; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — 130-nm albumin-bound paclitaxel; Gemcitabine

STUDY DESIGN:
Intervention Model Description: This is a single site, single-arm, open-label prospective clinical trial of the alternating GnP and mFOLFIRINOX regimens in selected patients with borderline-resectable pancreatic ductal adenocarcinoma (BR-PDAC) who have not received previous systemic or radiation therapy forPDAC.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Gemcitabine plus Nab-Paclitaxel and mFOLFIRINOX (Experimental): Patient has been diagnosed with borderline resectable pancreatic ductal adenocarcinoma (pancreatic cancer) and has not received systemic or radiation therapy. Treating physician has recommended neoadjuvant (pre-operative) chemotherapy and radiation, prior to surgery.
  Interventions: Drug: Nab-paclitaxel + Gemcitabine; Drug: modified FOLFIRINOX (mFOLFIRINOX)

INTERVENTIONS:
Drug: Nab-paclitaxel + Gemcitabine — Administered ion days 1, 8 and 15 of cycles 1 and 3 (28-day cycles).
Drug: modified FOLFIRINOX (mFOLFIRINOX) — Administered ion days 1 and 15 of cycles 2 and 4 (28-day cycles).

SUMMARY:
The purpose of this research is to study the effects and safety of alternating neoadjuvant chemotherapy on borderline resectable pancreatic cancer.

DETAILED DESCRIPTION:
Modified FOLFIRINOX (mFOLFIRINOX) and gemcitabine plus nab-paclitaxel (GnP) are two of the preferred chemotherapy treatments at this time. The U.S. Food and Drug Administration (FDA) has approved each of these treatments for patients with borderline resectable pancreatic cancer. This study will alternate these two neoadjuvant chemotherapy treatments (GnP and mFOLFIRINOX). The study doctors hope that alternating these treatments may improve the treatment response, improve tumor removal (also called "resectability"), and lower the risk of cancer coming back.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Diagnosis of BR-PDAC. The resectability should be officially determined with surgical oncologists at the Dartmouth Cancer Center (DCC) GI multidisciplinary Tumor Board based on NCCN Guidelines Version 2.2024 Pancreatic Adenocarcinoma.
* Patients must be able and willing to provide informed consent.
* Contrast-enhanced CT scan of the chest, abdomen, and pelvis performed within 45 days before registration.
* ECOG Performance Status: 0-1.
* Females of childbearing potential must have a negative pregnancy test done ≤ 14 days prior to study enrollment, and must agree to use a highly effective method of contraception throughout the course of protocol therapy.

Exclusion Criteria:

* Any prior receipt of chemotherapy or radiation therapy for PDAC.
* Known DPYD poor metabolizer genotype.
* Known BRCA1/2 or PALB2 mutations. If they are found to have BRCA1/2 or PALB2 mutation after inclusion to the trial, the participant will be taken off of protocol therapy (since platinum-containing therapy is preferred for these patients).
* Any confirmed second malignancy that is likely to require systemic therapy during the study period, in the opinion of the enrolling investigator.
* Any of the following baseline laboratory abnormalities:

  * Absolute neutrophil count (ANC) < 2,500/mm3
  * Platelet count < 100,000/mm3
  * Hemoglobin < 7 g/dL
  * Creatinine > 1.5 x upper limit of normal (ULN)
  * Total bilirubin > 1.5 x ULN
  * AST/ALT > 5 x ULN
* Any peripheral sensory neuropathy that meaningfully impairs performance of instrumental activities of daily living, as evaluated by the enrolling investigator.
* Patients who are unable to provide informed consent.
* Patients who are pregnant or breastfeeding.
* Patients who are incarcerated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-09-29 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2029-07-01 (Estimated)

PRIMARY OUTCOMES:
One-year event-free survival (1y-EFS) | I year
  One-year EFS is defined as completing one year from enrollment without the occurrence of any of the following events: 1) disease progression per Response Evaluation Criteria in Solid Tumors (RECIST), 2) surgery with R2 resection, 3) recurrent disease following surgery, or 4) death from any cause.

SECONDARY OUTCOMES:
Proportion of patients who complete the study intervention | 1 year
Proportion of patients who require dose modification | 1 year
Proportion of patients who undergo surgery | 1 year
Radiographic response (unconfirmed) after chemotherapy, per RECIST | 1 year
Surgical resection rate (R0, R1 and R2 resection) | 1 year
Pathologic response observed in the surgical specimen | 1 year
Recurrence-free survival (RFS) in patients who undergo surgery | 1 year
EFS (Event Free Survival) and OS (Overall Survival) | 1 year
Trend of CA19-9 | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States